CLINICAL TRIAL: NCT02641678
Title: Follow-up of Kryptogenic Stroke Patients With Implantable vs. Non-invasive Devices to Detect Atrial Fibrillation.
Acronym: TRACK-AF
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: TRACK-AF
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; stroke; implantable cardiac monitor; automated ECG analysis
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantation of cardiac monitor — In patients with kryptogenic stroke, a cardiac monitor was implanted to detect atrial fibrillation

SUMMARY:
Prospective mono-center diagnostic study determining potential discrepancies in identifying atrial fibrillation by intraindividually comparing different types of follow-up strategies:

1. How many stroke patients with atrial fibrillation are missed by standard stroke unit 24h- electrocardiography, and
2. what is the effectiveness of the extended invasive and non-invasive ECG analysis tools to detect atrial fibrillation in stroke patients?

DETAILED DESCRIPTION:
Atrial fibrillation often is paroxysmal and asymptomatic and, therefore, often not detected. Because atrial fibrillation is the leading risk factor for ischemic stroke, and oral anticoagulation is very efficacious for both primary and secondary stroke prevention in atrial fibrillation patients, detection of atrial fibrillation is essential to prevent stroke and stroke-induced disability and death. The incidence of atrial fibrillation and paroxysmal atrial fibrillation is particularly high in stroke patients. Short duration monitoring identified new atrial fibrillation in only about 5% to 10% of stroke patients. Estimates of missed paroxysmal atrial fibrillation in stroke patients go up to 40 000 patients in Germany per year.

Due to the known poor sensitivity of a 24h-ECG, all patients with stroke of unknown cause will undergo the above mentioned non-invasive and invasive ECG monitoring. Based on the data of these extended ECG-analyses, the rate of missed AF in conventionally diagnosed stroke unit patients could be determined by comparison to the 24h-ECG results. Additionally, a cost-benefit equation of the different ECG analysis tools will be calculated by comparison of the respective detection rates and the known follow-up costs.

Inclusion criteria: Patients years with acute ischemic stroke of unknown cause, monitored on a stroke unit undergoing routine diagnostic procedures (conventional 12-lead-ECG, 24h-ECG, echocardiography, cranial computed tomography or cranial magnetic resonance tomography, Transcranial Doppler and carotid duplex ultrasound, long-term blood pressure monitoring, standard laboratory investigations) Exclusion criteria: Stroke with known etiology, Stroke caused by intracranial hemorrhage

Diagnosis-as-usual:

- Standard 24h-ECG on stroke units according to existing guidelines

Investigational measure:

Non-invasive:

* Online ECG analysis during the standardized stroke unit- monitoring
* Ambulatory 7-day ECG monitoring

Invasive:

- atrial fibrillation detection by a permanently implantable direct cardiac rhythm monitor device in a period of up to 6 month

Duration of measures per patient:

2 weeks hospitalization, ~1 month rehabilitation, then implantation of the ECG device, and 6 months follow-up: 7.5 months in total

Primary outcome:

To determine the prevalence of undiagnosed AF in stroke patients undergoing the diagnostic standard (24h-ECG)

Secondary outcome:

Effectivity and cost-effectiveness ratios of the different ECG analyis tools

Description of the outcome:

Based on the obtained data, the prevalence of undiagnosed atrial fibrillation in stroke patients whom atrial fibrillation is missed by the standard diagnostic procedure (24h-ECG) will be determined by different extensive non-invasive and invasive ECG monitoring tools.

Additionally, following values of the applied ECG analysis tools will be calculated and compared:

* Sensitivity: (true positives) / (true positives + false negatives)
* Specificity: (true negatives) / (true negatives + false positives)
* Positive predicted value: (true positives) / (true positives + false positives)
* Negative predicted value: (true negatives) / (true negatives + false negatives)

Safety:

The implantable direct cardiac rhythm monitor device is an established and widely used diagnostic procedure in patients with unexplained syncope.

ELIGIBILITY:
Inclusion Criteria:

Patients years with acute ischemic stroke of unknown cause, monitored on a stroke unit undergoing routine diagnostic procedures (conventional 12-lead-ECG, 24h-ECG, echocardiography, cCT or cMRI, Transcranial Doppler and carotid duplex ultrasound, long-term blood pressure monitoring, standard laboratory investigations)

Exclusion Criteria:

* Stroke with known etiology, Stroke caused by intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke of unknown etiology
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of undiagnosed AF in stroke patients undergoing the diagnostic standard (24h-ECG) | 7.5 months
  Based on the obtained data, the prevalence (in percent) of undiagnosed AF in stroke patients whom AF is missed by the standard diagnostic procedure (24h-ECG) will be determined by different extensive non-invasive and invasive ECG monitoring tools

SECONDARY OUTCOMES:
Diagnostic accuracy of the automated software based ECG analysis in comparison to the "gold-standard" the implanted cardiac monitor | 7.5 months
  The Sensitivity (in percent), the Specificity (in percent), the positive predictive value (in percent) and the negative predictive value (in percent) will be calculated for the automated ECG software analysis in comparison to the "gold-standard" the implanted cardiac monitor

OTHER OUTCOMES:
Diagnostic accuracy of the automated software based ECG analysis in comparison to the standard methods (routine ECG, 24h longterm ECG) | 7.5 months
  The Sensitivity (in percent), the Specificity (in percent), the positive predictive value (in percent) and the negative predictive value (in percent) will be calculated for the automated ECG software analysis in comparison to the actual diagnostic standard the routinely performed ECG+longterm ECG.
Cost efficacy of the different methods (automated software based ECG analysis and implantable cardiac monitor) | 7.5 months
  The data can be helpful to increase the cost efficacy. There are 3 hypotheses. 1.) The software analysis is reliable enough to detect AF than an implantable device is no longer needed.
  2.) The software analysis is unreliable 3.) The software analysis has a high negative predictive value and can provide as a preselection tool. Patients with probable AF calculated by the software analysis have a higher profit by the implantation than the patient with no AF calculated by the software.

CONTACTS AND LOCATIONS:
Overall Officials: Dittrich Ralf, MD, Principal Investigator — Department of Neurology, University of Muenster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bettin M, Dechering D, Kochhauser S, Bode N, Eckardt L, Frommeyer G, Reinke F. Extended ECG monitoring with an implantable loop recorder in patients with cryptogenic stroke: time schedule, reasons for explantation and incidental findings (results from the TRACK-AF trial). Clin Res Cardiol. 2019 Mar;108(3):309-314. doi: 10.1007/s00392-018-1358-4. Epub 2018 Aug 22. PMID 30167809
- [Derived] Reinke F, Bettin M, Ross LS, Kochhauser S, Kleffner I, Ritter M, Minnerup J, Dechering D, Eckardt L, Dittrich R. Refinement of detecting atrial fibrillation in stroke patients: results from the TRACK-AF Study. Eur J Neurol. 2018 Apr;25(4):631-636. doi: 10.1111/ene.13538. Epub 2018 Feb 13. PMID 29205690